CLINICAL TRIAL: NCT06651008
Title: The New Factors That Lead to Conversion Surgery in Patients with Duodenal Perforation When Initial Conservative Therapy is Not Completed
Brief Title: The New Transition Factors to Surgery of Duodenal Perforation
Status: Completed | Type: Observational
Sponsor: Toho University (Other)
Responsible Party: Principal Investigator, Kenjiro Ishii, MD. PhD, lecturer, head of upper gastrointestinal surgery group of toho ohashi hospital, Toho University
Other Study IDs: Toho-retrospective study 1
Record Dates: First submitted 2024-10-15; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Duodenum Ulcer Perforation
Keywords: conversion to surgery; conservative management,

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Conservative treatment completed group: The groupthat completed the conservative treatment for dudenum perforation.
- Conversion to surgery group: The group that needed conversion to surgery for duodenum perforation.

SUMMARY:
In this study,investigators sought to identify new transition factors in the initial evaluation of cases requiring conversion to surgery for duodenal ulcer perforation.

This was a retrospective study performed at investigators' hospital between January 2012 and July 2023 with upper gastrointestinal perforation. 27 patients, who underwent conservative management for the duodenal ulcer perforation, were extracted. Investigators researched the transition rate to surgery and the following factors: 1. Patient background, 2. Time from onset to hospital visit, 3. Vital signs and inflammatory findings on arrival, 4. CT findings of duodenal ulcer perforation and degree / shape of liver coverage for the perforation, and the extent of ascites.

ELIGIBILITY:
Inclusion Criteria:

* patients of upper gastrointestinal perforation

Exclusion Criteria:

* DNR patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This was a retrospective study performed at our hospital between January 2012 and July 2023 with upper gastrointestinal perforation, and included 74 patients admitted to our hospital.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
The rate of conversion to surgery from conservative management for duodenal ulcer perforation. | nearly within 3days
  Th investigators reasearched the transition rate to surgery based on the following factors: 1. Patient background, 2. Time from onset to hospital visit, 3. Vital signs and inflammatory findings on arrival, 4. CT findings of duodenal ulcer perforation and degree / shape of liver coverage for the perforation, and the extent of ascites.

IPD SHARING:
Plan to Share IPD: Yes
Imaging findings etc of study patients will be provided in an anonymous form.
Supporting Information: Study Protocol
Time Frame: almost 1 year